CLINICAL TRIAL: NCT03505658
Title: Abriendo Caminos 2: Clearing the Path to Hispanic Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: California State University, Fresno Foundation (Other); Iowa State University (Other); University of Houston (Other); University of Puerto Rico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15503
Record Dates: First submitted 2018-02-01; First posted 2018-04-23 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Obesity; Childhood Obesity; Nutrient; Excess; Community Health Education
MeSH Terms: conditions — Obesity; Pediatric Obesity; Health Education | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The Intervention is educational with 6 workshops for 2 hrs a week. Data/ assessments are collected, pre and post the 6 weeks intervention and 6 months post follow-up.
  Interventions: Behavioral: Education and Behavior
- Control (No Intervention): One or two non-intervention related workshop talks are given; 1 hr each during the same 6 weeks as the intervention arm. Pre and post assessment/ data collection and 6 months follow-up are completed.

INTERVENTIONS:
Behavioral: Education and Behavior — Involves 6-weeks of education related to healthy behaviors, nutrition, and exercise.
  Arms: Intervention

SUMMARY:
Obesity is significantly higher in specific ethnic groups and, in particular, Hispanics. There is an urgent need to implement culturally-sensitive lifestyle interventions and educational programs to decrease the burden of obesity and obesity-related metabolic diseases in Hispanic populations. Accordingly, our overreaching goal is to tailor an existing and successful community-based program, Abriendo Caminos, to leverage effectiveness in promoting healthy nutrition and life-style behaviors among low income, low literacy Hispanic-heritage families. Our multi-function integrated project proposes to (a) adapt Abriendo Caminos for 6-18 year-old children from Mexican and Puerto Rican heritage in five different locations (California, Illinois, Iowa, Puerto Rico, and Texas) and (b) Train existing professionals (in Extension and community agencies) and future professionals (Hispanic university students) to meet the specific needs of this population. Our central hypothesis is that participation in a 6-week community-based program will prevent childhood obesity/maintain healthy weight by significantly increasing: (a) healthy dietary behavior patterns and basic knowledge of nutrition; (b) physical activity levels; and (c) the organization of collective/shared family mealtimes. The implementation of this culturally sensitive, workshop-based curriculum in different regions across the country will help to train the next generation of professionals in Extension and communities to deliver programs that meet the needs of Hispanic families. The integration of Hispanic college students in program implementation via an experiential learning course will further strengthen the program, as well as increase recruitment and retention of Hispanic students, increasing the capacity of Hispanic communities to meet their own needs in the future.

ELIGIBILITY:
Inclusion Criteria:

* a family member being 6-18 years of age
* at least 1 parent being of Hispanic-heritage from Mexican or Puerto Rican origin

Exclusion Criteria:

* no child in the age range of 6-18 years of age
* No parents being of Hispanic-heritage from Mexican or Puerto Rican origin

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-04-10 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
BMI | Baseline
  Body mass index = weight per height square in metrics
BMI | 6-month post intervention
  Body mass index = weight per height square in metrics

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - California State University, Fresno, California
  - University of Illinois at Urbana-Champaign, Urbana, Illinois
  - Iowa State University, Ames, Iowa
  - University of Houston, Houston, Texas
- University of Puerto Rico, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided
If researchers are interested in obtaining study data please contact the PI for further discussions and what approvals such as IRB is needed to gain access to deidentified data.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-04-06): https://cdn.clinicaltrials.gov/large-docs/58/NCT03505658/SAP_000.pdf
  • Study Protocol (2018-04-06): https://cdn.clinicaltrials.gov/large-docs/58/NCT03505658/Prot_001.pdf